CLINICAL TRIAL: NCT02668315
Title: A Phase I-II Open-label Study of UM171 Expanded Cord Blood in a Fed-batch Culture System (UFCB-001) in Patients Who Need an Allogeneic Hematopoietic Stem Cell Transplant But Lack a Suitable Donor
Brief Title: Expanded Cord Blood in Patients in Need of an Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Hopital de l'Enfant-Jesus (Other); Vancouver General Hospital (Other); St. Justine's Hospital (Other); Stem Cell Network (Other)
Responsible Party: Principal Investigator, Sandra Cohen, MD, Maisonneuve-Rosemont Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UM0128171
Record Dates: First submitted 2016-01-15; First posted 2016-01-29 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Intervention name: Transplantation of cord blood expanded with UM171 Prethaw CB cell count prior to manipulation: CD34+ cell count 1.0-4.9 x 10E5/kg and TNC superior or equal to 2.0 x 10E7/kg
  Interventions: Biological: Transplantation of cord blood expanded with UM171
- Cohort 2 (Experimental): Intervention name: Transplantation of cord blood expanded with UM171 Prethaw CB cell count prior to manipulation: CD34+ cell count 0.5-4.9 x 10E5/kg and TNC superior or equal to 1.5 x 10E7/kg
  Interventions: Biological: Transplantation of cord blood expanded with UM171
- Cohort 3 (Experimental): Intervention name: Transplantation of cord blood expanded with UM171 Prethaw CB cell count prior to manipulation: CD34+ cell count 0.25-4.9 x 10E5/kg and TNC superior or equal to 1.25 x 10E7/kg
  Interventions: Biological: Transplantation of cord blood expanded with UM171

INTERVENTIONS:
Biological: Transplantation of cord blood expanded with UM171 — Myeloablative or submyeloablative conditioning regimen followed by an expanded cord blood transplant

SUMMARY:
Allogeneic hematopoietic stem cell transplantation is a life-saving procedure in patients with blood cancers, but only 25% of transplant candidates have a sibling donor. A matched unrelated donor can be found for 60% of patients but this number is lower for non-Caucasians. Cord blood (CB), another source of stem cells, has major advantages over unrelated donors including immediate availability, better permissiveness in immune mismatches between donor and transplant recipient, better availability for non-Caucasians, and less graft versus host disease, a complication frequently seen after transplant which negatively affects quality of life. Unfortunately, the use of CB is still limited in adults because of the small number of stem cells. UM171, a molecule with hematopoietic stem cell expansion properties, has been shown to increase cord blood stem cells 13 fold. In this trial, Investigators will use UM171 treated CB in patients who need a transplant but lack an acceptable donor.This protocol seeks to test the safety of CB cells expanded with UM171, and to determine the kinetics of engraftment as well as the minimal cord blood unit cell dose that when expanded achieves prompt engraftment.

DETAILED DESCRIPTION:
Investigators are proposing a phase I-II, Canadian multi-center, open-label study of UM171 ex vivo expanded CB transplant in 25 patients who need an allogeneic hematopoietic stem cell transplantation (HSCT) but lack a Human Leucocyte Antigen (HLA) matched donor.

Investigators key primary and secondary objectives include:

1. To establish the feasibility of expanding cord blood units for allogeneic cord blood transplantation.
2. To establish the safety and identify unexpected toxicities associated with the transplantation of cord blood cells expanded with UM171/fed-batch culture system.
3. To measure kinetics of neutrophil and platelet recovery.
4. To determine minimal cord blood unit cell dose (Total Nucleated Cell (TNC)/CD34+ cells) that when expanded achieves prompt engraftment as a single cord transplant.

Methodology:

Patients with a hematologic malignancy and an indication for allogeneic HSCT who lack a matched unrelated donor will receive a myeloablative or submyeloablative conditioning regimen followed by infusion of UM171 expanded CB graft. Accrual is expected to last 18 months and patients will be followed for 3 years.

Expected benefits:

Investigators expect that expansion with UM171/fed-batch will be safe and lead to both rapid and sustained engraftment. This will likely decrease the high early morbidity/mortality of CB HSCT and improve access to transplant, especially ethnic minorities. In addition, if low cell dose is solved, patients will benefit from CB's lower risk of chronic (graft versus host disease) GVHD, a major cause of morbidity.

.

ELIGIBILITY:
Inclusion

1. 3-64 years old (Pediatric patients will become eligible only after 5 adult patients have been enrolled in the study and received the UM171 expanded product).
2. Weight ≥ 12kg
3. Underlying hematologic malignancy excluding primary myelofibrosis requiring an unrelated donor allogeneic HSC transplant (as defined by the transplant center) but patient lacks an 8/8 HLA identical donor or disease requires an urgent transplant and cannot wait the required time to identify an unrelated donor.
4. Availability of at least 3 cord bloods with HLA match ≥ 4/6 and ≥4/8 and meeting the following requirements:

   * CB to be expanded: CD34+ cell count 1.0-4.9 x 10E5/kg for cohort 1, 0.5-4.9 x 10E5/kg for cohort 2, and 0.25-4.9 x 10E5/kg for cohort 3; nucleated cell count ≥ 2.0 x 10E7/kg for cohort 1, ≥ 1.5 x 10E7/kg for cohort 2, and ≥ 1.25 x 10E7/kg for cohort 3.
   * Non expanded cord: TNC count ≥ 2.0 x 10E7/kg with CD34 min of 1 x 10E5/kg or minimum of 1.5 x 10E7 TNC/kg with 1.8 x 10E5 CD34+ cells/kg.
   * Back up cord: TNC count ≥ 1.5 x 10E7/kg with CD34 min of 1 x 10E5/kg
5. Left ventricular ejection fraction > 40%.
6. Karnofsky score ≥ 70%
7. Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and diffusing capacity corrected for hemoglobin (DLCOc) ≥ 50% of predicted
8. Bilirubin < 2 x upper limit of normal (ULN) unless felt to be related to Gilbert's disease or hemolysis; AST (aspartate aminotransferase) and ALT (alanine aminotransférase) ≤ 2.5 x ULN; alkaline phosphatase ≤ 5 x ULN.
9. Measured or estimated creatinine clearance ≥ 60 ml/min/1.73m2.

Exclusion

1. Myeloablative transplant within 24 months.
2. Uncontrolled infection.
3. Presence of a malignancy other than the one for which the UCB transplant is being performed and the expected survival related to the malignancy is estimated to be less than 75% at 5 years.
4. HIV positivity.
5. Hepatitis B or C infection with measurable viral load.
6. Liver cirrhosis.
7. Availability of a cord with ≥ 5 x 105/kg CD34+ cells.
8. Pregnancy, breastfeeding or unwillingness to use appropriate contraception.
9. Participation in a trial with an investigational agent within 30 days prior to entry in the study.
10. Patient unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and tests.
11. Any abnormal condition or laboratory result that is considered by the principal investigator capable of altering patient condition or study outcome.

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Monitoring adverse events, toxicities and medical evolution | up to 36 months post transplant
  To identify unexpected toxicities associated with transplantation using cord blood cells expanded with UM171/fed-batch culture system by means of history, physical examination and laboratory evaluation. All adverse events will be evaluated for duration, intensity, and causal relationship with the study medication and followed to the end of the study or until resolution.

SECONDARY OUTCOMES:
Feasibility of cord blood expansion using UM171 (transplant success) | 18 months
  The feasibility of expanding cord blood units for allogeneic cord blood transplantation in adults will be evaluated by determining the percentage of selected grafts that will be successfully expanded in the absence of technical hurdles such as contamination or unexpected technical failure, and that will meet release criteria and be successfully infused in patients.
Kinetics of hematopoietic recovery | 42 days post transplant
  Time to neutrophil engraftment is defined as the first day of attainment of an absolute neutrophil count (ANC) ≥ 0.5 x 109/L for 3 consecutive days as per Center for International Blood and Marrow Transplant Research (CIBMTR) standards.
  Platelet engraftment is defined as the first day of a sustained platelet count ≥ 20 x 109/L with no platelet transfusion in the preceding 7 days as per CIBMTR standards.
Minimal cord blood cell dose that when expanded achieves prompt engraftment | up to 12 months
  The minimal cord blood unit cell dose (TNC/CD34+) that, once expanded, achieves prompt engraftment as a single cord transplant will be defined as the lower cord blood cell dose that satisfies all of the following conditions for umbilical cord blood (UCB) dose reduction , i.e.:
  * Minimum of 3 patients who will have received a single cord transplant (no back-up cord),
  * Cord to be expanded contains less than 2.0 x 105 CD34+/kg at thaw pre-expansion in cohort 1 and less than 1.0 x 105 CD34+/kg at thaw pre-expansion in cohort 2
  * Engraftment must have occurred within 18 days.
Correlation between neutrophil and platelet engraftment and CD34+ and CD34+CD45RA- dose | 42 days post transplant
  Time to neutrophil and platelet engraftment will be correlated to the CD34+ and the CD34+CD45RA- dose (which includes all human hematopoietic stem cells (HSCs): long term and short term repopulating cells) contained in the expanded graft. Expansion and cultures might change the characteristics and behaviour of CD34+ cells, hence the need to look at the correlation between primitive CD34+CD45RA- subpopulation and engraftment.
Incidence of primary and late graft failure | 42 days post transplant
  The patient will be declared as having developed primary graft failure if:
  * Lack of neutrophil engraftment by day 42.
  * Infusing another stem cell source prior to day 42 (other than the nonmanipulated cord and back up cord).
  * < 5% donor chimerism after day +14 up to and including day +42 after transplant.
  * Death from day 28 to 42 without neutrophil engraftment.
  Secondary or late graft failure when:
  • ANC drops below 0.5 x 109/L for 14 consecutive days unresponsive to growth colony stimulating factor (G-CSF) witout identifiable cause (medication, viral infection, vitamin deficience or other)
Incidence of backup cord infusion and graft dominance | 7, 14, 21, 28, 56, 100 days and at 6 and 12 months
  This evaluation will be performed in lymphoid and myeloid cells to determine the expanded cord's role in short and long term engraftment in patients. Cell sorting to examine chimerism of different cell subsets will be performed with complex of differentiation (CD) such as CD3, CD33, CD56, CD14 and CD19 to determine the proportions in which donor's immune cells are represented in the graft recipient.
  Donor cell engraftment is defined as donor cell (lymphoid or myeloid) chimerism ≥ 5% by day +42 post transplant. Full donor chimerism is defined as ≥ 95% donor myeloid and lymphoid chimerism.
Incidence of acute and chronic GVHD | through study completion (3 years follow-up)
  The incidence of acute and chronic GVHD will be evaluated throughout the study using NIH criteria. Acute GVHD will be defined as classic acute (time of onset of symptoms ≤ 100 days) or persistent, recurrent, or late onset acute GVHD (time of onset of symptoms > 100 days) as defined by the NIH.
  Patients will be assessed for the presence of chronic GVHD at each medical evaluation. Data will be collected directly from providers and chart review according to the recommendations of the NIH Consensus Conference.
Incidence of severe infectious complications | through study completion (3 years follow-up)
  any grade 3 infection will be tabulated as well as any of the following infections requiring systemic therapy will be captured: invasive candidiasis, aspergillus, other invasive fungi, cytomegalovirus (CMV), adenovirus, Epstein-Barr virus (EBV), Human herpes virus (HHV-6), herpes simplex (HSV), varicella-zoster virus (VZV), Pneumocystis carinii pneumonitis (PCP), toxoplasmosis and mycobacterium. Severity of infections will be graded according to the Technical Manual of Procedure of the Blood and Marrow Transplant Clinical Trials Network.
T cell evaluation (Cluster of differentiation (CD) 4+ and CD8+) | 3, 6, 12, and 18 months
  Multiparametric flow cytometry to quantify the proportion of naïve (CD45RA+/CD27+) and memory (CD45RA-/CD27+) cells.
B cell evaluation | 3, 6, 12, and 18 months
  The outcome (success or failure) in B cell recovery will be evaluated by flow cytometry, immunoglobulin measurements and PCR for donor cell chimerism.
Natural Killer (NK) cell evaluation | 3, 6, 12, and 18 months
  The outcome (success or failure) in NK cell recovery will be evaluated by flow cytometry and PCR for donor cell chimerism.
Transplant related mortality (TRM) | 100 days and 1,2, 3 years post transplant
  Incidence of TRM will be monitored throughout the study and in particular at 100 days, 1, 2, and 3 years post transplantation. If it should exceed 30% at day 100, stopping rules may apply that could prematurely terminate the trial.
progression free survival | 100 days an 1,2, 3 years post transplant
  Progression free survival (PFS) will be monitored throughout the study and in particular at 1, 2, and 3 years post-transplant.
  PFS will be measured from time of transplant until progression, death or last follow-up.
  PFS: an event is defined as relapse/progression or death.
Overall survival | 100 days an 1,2, 3 years post transplant
  Overall survival (OS) will be monitored throughout the study and in particular at 1, 2, and 3 years post-transplant.
  OS will be measured from time of transplant until progression, death or last follow-up.
  OS: an event is defined as death.
Incidence of engraftment syndrome requiring therapy | 24 hours post transplant and during follow-up (3 years)
  Patients will be monitored for the occurrence of engraftment and preengraftment syndromes (ES and PES) as well as the necessity for treatment. Diagnostic criteria for ES are noninfectious fever plus any of the following: skin rash, pulmonary infiltrates, hepatic dysfunction, or diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Cohen, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu B, Klatt D, Zhou Y, Manis JP, Sauvageau G, Pellin D, Brendel C, Williams DA. UM171 enhances fitness and engraftment of gene-modified hematopoietic stem cells from patients with sickle cell disease. Blood Adv. 2024 Nov 26;8(22):5885-5895. doi: 10.1182/bloodadvances.2024013932. PMID 39293082
- [Derived] Cohen S, Bambace N, Ahmad I, Roy J, Tang X, Zhang MJ, Burns L, Barabe F, Bernard L, Delisle JS, Kiss T, Lachance S, Roy DC, Veilleux O, Sauvageau G. Improved outcomes of UM171-expanded cord blood transplantation compared with other graft sources: real-world evidence. Blood Adv. 2023 Oct 10;7(19):5717-5726. doi: 10.1182/bloodadvances.2023010599. PMID 37467030
- [Derived] Dumont-Lagace M, Li Q, Tanguay M, Chagraoui J, Kientega T, Cardin GB, Brasey A, Trofimov A, Carli C, Ahmad I, Bambace NM, Bernard L, Kiss TL, Roy J, Roy DC, Lemieux S, Perreault C, Rodier F, Dufresne SF, Busque L, Lachance S, Sauvageau G, Cohen S, Delisle JS. UM171-Expanded Cord Blood Transplants Support Robust T Cell Reconstitution with Low Rates of Severe Infections. Transplant Cell Ther. 2021 Jan;27(1):76.e1-76.e9. doi: 10.1016/j.bbmt.2020.09.031. Epub 2020 Oct 3. PMID 33022376
- [Derived] Cohen S, Roy J, Lachance S, Delisle JS, Marinier A, Busque L, Roy DC, Barabe F, Ahmad I, Bambace N, Bernard L, Kiss T, Bouchard P, Caudrelier P, Landais S, Larochelle F, Chagraoui J, Lehnertz B, Corneau S, Tomellini E, van Kampen JJA, Cornelissen JJ, Dumont-Lagace M, Tanguay M, Li Q, Lemieux S, Zandstra PW, Sauvageau G. Hematopoietic stem cell transplantation using single UM171-expanded cord blood: a single-arm, phase 1-2 safety and feasibility study. Lancet Haematol. 2020 Feb;7(2):e134-e145. doi: 10.1016/S2352-3026(19)30202-9. Epub 2019 Nov 6. PMID 31704264